CLINICAL TRIAL: NCT04773236
Title: Evaluation of Buffered Local Anesthesia in Dental Extraction: A Randomized Clinical Study.
Brief Title: Evaluation of Buffered Local Anesthesia in Dental Extraction.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Danny Benjamin, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 206120
Record Dates: First submitted 2021-02-21; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Buffered Local anesthesia (Active Comparator): Sodium bicarbonate with 2% lidocaine and 1:80.000 epinphrine
  Interventions: Drug: sodium bicarbonate 8.4%; Device: Mixing pen (onset buffering system)
- Non Buffered Local anesthesia (Placebo Comparator): 2%lidocaine with 1:80.000 epinphrine.
  Interventions: Drug: 2%lidocaine with 1:80.000 epinphrine

INTERVENTIONS:
Drug: sodium bicarbonate 8.4% — mixing the sodium bicarbonate with 2%lidocaine and 1:80.000 epinphrine using mixing pen (onset buffering system)
  Arms: Buffered Local anesthesia
Drug: 2%lidocaine with 1:80.000 epinphrine — injection
  Arms: Non Buffered Local anesthesia
Device: Mixing pen (onset buffering system) — Premixing of the two solutions sodium bicarbonate and lidocaine with epinphrine before the local anesthesia adminstration to the patient
  Arms: Buffered Local anesthesia

SUMMARY:
To compare pain during injection, onset of anesthesia and effectiveness of anesthesia using buffered versus non- buffered 2% lidocaine with 1:80,000 adrenaline in dental extraction.

DETAILED DESCRIPTION:
The investigators will conduct a prospective, randomized, single-blinded study, the sample will include 100 patients (extraction) who need dental extraction of upper teeth (premolar and molar teeth). The predictor variable is the use of buffered 2% lidocaine with 1:80,000 adrenaline and non-buffered 2% lidocaine with 1:80,000 adrenaline. The patients will be randomly assigned into two groups of 50 patients each using Microsoft Excel 2016; the first group (study group) will undergo dental extraction after receiving buffered 2% lidocaine with 1:80,000 adrenaline, the second group (control group) will undergo dental extraction after receiving non-buffered 2% lidocaine with 1:80,000 adrenaline. The outcome variables include pain during injection, onset of anesthesia and effectiveness of anesthesia on buffered and non-buffered group.

ELIGIBILITY:
Inclusion Criteria:

1. Give written, informed consent (both the subject and the legal guardian).
2. Be 18-65 years of age. 3.Be able to comprehend the visual analog scale (instructions given to ascertain this).

4.Be able to comprehend the verbal rating scale (instructions given to ascertain this).

5.upper premolars and molars extraction.

Exclusion Criteria:

1. Patient under 18 years.
2. pregnant women.
3. patient with uncontrolled systemic disease that are contraindicated for dental extraction. 4- patient taking medication that interfere with the assessment of local anesthetic such as narcotics and antidepressants .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-22 (Estimated); Primary Completion 2021-05-22 (Estimated); Study Completion 2021-08-22 (Estimated)

PRIMARY OUTCOMES:
Pain during Injection | Immediately after Injection
  Numerical rating scale from 0-10 that (0) mean no pain and (10) worst pain
Onset of anesthesia | 30 seconds to 90 seconds
  probing marginal gingiva
Effectiveness of anesthesia | during procedure
  number of carpules used